CLINICAL TRIAL: NCT01412086
Title: Inter-rater and Intra-rater Reliability of the Global Eyebrow Assessment Scale
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 192024-068
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Healthy volunteers. No treatment (intervention) was received.
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — No Intervention.

SUMMARY:
This study evaluated the inter- and intra-rater reliability of the GEBA Scale with photonumeric guide for the assessment of overall eyebrow fullness. There is no treatment (intervention) associated with this study.

ELIGIBILITY:
Inclusion Criteria:

* Willing to remove makeup and jewelry at each visit
* Willing to have photographs taken of the facial area

Exclusion Criteria:

* Permanent eyebrow makeup (i.e., tattooing) or eyebrow implants of any kind
* Eyebrow extension application within 3 months of study entry
* Eyebrow tint or dye application within 2 months of study entry
* Eyebrow grooming (i.e., tweezing, waxing, or threading) between visits that is not part of the current routine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 112
Completed | 112
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 112
Age Continuous [Mean (Full Range); unit: Years] | 44.3 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Reliability of Physician Raters Using the Global Eyebrow Assessment (GEBA) Scale
Description: Inter-rater agreement (among raters) of the GEBA scores (1=very sparse, 2=sparse, 3=full, 4=very full) to assess eyebrow fullness was evaluated using Kendall's coefficient of concordance (Kendall's W). Each of 7 raters scored 112 subjects' eyebrows using the GEBA Scale at 2 different time points at day 1. The overall inter-rater agreement for Kendall's W for all raters combined was estimated based on the average of the scores from those 2 different time points. The degree of agreement of the point estimates of Kendall's W was interpreted according to the reference range scale that was pre-defined as: ≤ 0: poor, 0.00-0.20: slightly, 0.21-0.40: fair, 0.41-0.60: moderate, 0.61-0.80: substantial and 0.81-1:00: almost perfect. The 95% confidence interval for Kendall's W was provided.
Time Frame: Day 1
Measure: Number (95% Confidence Interval); unit: Kendall's W
Arm/Group | All Participants
Number analyzed (Participants) | 112
Kendall's W | 0.889 [0.695 to 1.000]

2. Primary Outcome: Intra-rater Reliability of Physician Raters Using the Global Eyebrow Assessment (GEBA) Scale
Description: Intra-rater (within raters) agreement of the GEBA scores (1=very sparse, 2=sparse, 3=full, 4=very full) to assess eyebrow fullness was evaluated by weighted Kappa statistics. Weighted Kappa statistics were calculated for each of 7 raters who evaluated 112 subjects using GEBA scale, assessing agreement between 2 different time points at day 1. The overall intra-rater agreement for Kappa statistics for all raters combined was estimated by pooling Kappa statistics for each rater using a chi-square statistic. The degree of agreement of the point estimates of Kappa statistics was interpreted according to the reference range scale that was predefined as: ≤ 0: poor, 0.00-0.20: slightly, 0.21-0.40: fair, 0.41-0.60: moderate, 0.61-0.80: substantial and 0.81-1:00: almost perfect. The 95% confidence interval for Kappa statistics was provided.
Time Frame: Day 1
Population: All enrolled participants.
Measure: Number (95% Confidence Interval); unit: Kappa statistics
Arm/Group | All Participants
Number analyzed (Participants) | 112
Kappa statistics | 0.807 [0.780 to 0.834]

ADVERSE EVENTS:
Description: Adverse event data were not collected/assessed.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.